CLINICAL TRIAL: NCT04695912
Title: The Effect of Accelerometer Guided App Feedback on Change in Activity in Patients With Low Back Pain
Brief Title: The Effect of Accelerometer Guided App Feedback on Change in Activity in Patients With Low Back
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Anna Katrine Skovsgaard Itenov, senior registrar, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H-17010038
Record Dates: First submitted 2020-12-08; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Low Back Pain; Radiculopathy Lumbar; Sciatica
MeSH Terms: conditions — Low Back Pain; Sciatica

STUDY DESIGN:
Intervention Model Description: crossover, open-label, randomized, controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Initial activity tracker with feedback followed by control period (Other): Initial activity tracker with feedback followed by control period
  Interventions: Device: The SENS motion® sensor
- Initial control period followed by activity tracker with feedback (Other): Initial control period followed by activity tracker with feedback
  Interventions: Device: The SENS motion® sensor

INTERVENTIONS:
Device: The SENS motion® sensor — The sensor is a wearable physical tracker giving investigators feedback about daily activity
  The SENS motion® system consists of:
  The sensor 'SENS Motion Patch' A smart-phone application 'SENS motion´
  SENS motion cloud storage database, a web-based visualization of data for the healthcare team
  The iSpine app shows activity-information recorded by the sensor to the patient and gives nudges to activity.
  Other Names: iSpine app (InterMedCon)

SUMMARY:
In a cross-over, open-label, randomized, controlled trial, the investigators aim to determine if the daily activity level in patients with LBP can be increased via feedback from an app, connected to a wearable sensor of physical activity.

DETAILED DESCRIPTION:
The aim of the study is to determine if a wearable device that measure physical activity and a smartphone application with nudges and feedback increase the physical activity level of patients with low back pain over a 14 days period.

Secondary to determine how many of the patients, that use the smartphone application, and if they perceived the feedback as inspiring.

And to explore, if a potential effect of the device and smartphone application depended on the baseline activity level, gender, diagnoses, age, education level and previous exercise experience.

1. Is there a difference in average (mean) daily number of active minutes (defined as walking, cycling, running or exercise) over the 14 days intervention period compared to the 14 days control period.
2. If there is an effect of the device and smartphone application, then determine how many of the patients, that use the smartphone application, and if they perceived the feedback as inspiring.

   To explore, if a potential effect of the device and smartphone application depended on the baseline activity level, gender, diagnoses, age, education level and previous exercise experience.
3. Is the outcome measures; function measured by sensor, the subjective measurements as pain, stiffness and function, responsive to the intervention compared, to the global scale. 4. Is the patient´s self-evaluated change in activity in the intervention period compared to the baseline period and the control period corelated to the changes in activity measured by the sensor.

The investigators will make a Cross-over, randomized, open label, controlled trial.

Patients will be included from the outpatient clinic, The Department of Rheumatology, Rigshospitalet - Glostrup, Region Hovedstaden, Denmark Inclusions criteria

* Aged 18 years or older
* Non-specific low back pain, spinal stenosis or radiculopathy.
* Not referred for surgical evaluation.
* Patients who scored ≥ 20 point at the Oswestry Disability Index Exclusion criteria
* Patients with comorbidity that prevent them for participating in the study.
* Patients who are judge by the principal investigator to not speak Danish sufficiently to enable them to comprehend the study information and app feedback.
* Patients who already monitor their activity by a watch, on a daily basis.
* Patients with allergy for band aid
* Patients who are pregnant or breastfeeding

The patients are randomized to start with intervention + standard-of-care or only standard-of-care. After completion of the first period the patients will cross-over to the other period.

The patients are randomized by closed envelope. Using a randomization list from randomization.com.

Intervention period

The patients wear the SENS motion patch for 14 days and received daily updates on activity, and suggestions for improvements. During the intervention period the patients receive standard-of-care.

Control period

The patients wear the SENS motion patch for 14 days, but do not receive any feedback from the sensor. During the control period the patients receive standard-of-care.

Standard-of-care

At the outpatient clinic patients are examined by a doctor, receive a diagnosis and may undergo MRI to identify other causes for back pain. They are not offered any training program at the hospital, but they are recommended to stay active and exercise. Some may have a consultation with a physiotherapist one to two times who repeat the advice. Patients are informed that despite pain, they cannot harm their spine by work, exercise or performing daily activities, and that medical staff do not discourage any activities.

Name of the investigational device

SENS motion®, SENS-Innovation ApS

Titangade 11, 2. - 2200 Kbh. N.

Sensor

The SENS motion® system consists of:

* The sensor 'SENS Motion Patch'
* A smart-phone application 'SENS motion´

  * SENS motion cloud storage database, a web-based visualization of data for the healthcare team

ELIGIBILITY:
Inclusion Criteria:

* non-specific low back pain, spinal stenosis, radiculopathy
* moderate disability or worse (20-100 points on Oswestry Disability Index)

Exclusion Criteria:

* co-morbidity making the patients unable to move
* unsufficient Danish-skills
* patients who already monitored their activity by watch or phone on a daily basis
* allergy to band-aid
* pregnancy or breast-feeding
* patients referred for back-surgical evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Average daily activity | 1 month
  The Primary outcome was defined as the difference in average (mean) daily number of minutes in activity (defined as the sum of time spent with standing, walking, cycling and exercising) in 14 days intervention period compared to 14 days control period, registered by the sensor.

CONTACTS AND LOCATIONS:
Overall Officials: Anna katrine Itenov, MD, Principal Investigator — COPEBACK, Rigshospitalet
Locations (1):
- COPEBACK, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No